CLINICAL TRIAL: NCT03368313
Title: Non-elastic Compression Garment Therapy Versus Control for Deep Vein Thrombosis: A Bayesian Adaptive Randomized Trial
Brief Title: Non-elastic Compression Garment Therapy Versus Control for Deep Vein Thrombosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pró Circulação® (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Circaid
Record Dates: First submitted 2017-11-28; First posted 2017-12-11 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2021-09

CONDITIONS: Deep Vein Thrombosis; Post Thrombotic Syndrome
Keywords: Nonelastic compression theraphy; Compression theraphy; Compression stockings
MeSH Terms: conditions — Venous Thrombosis; Postthrombotic Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Compression arm (Experimental): The compression arm will receive an adjustable velcro compression device for the calf (Circaid Juxtalite® Lower Leg; Medi Gmbh, Bayreuth, Germany), thigh and knee (Circaid Juxtafit; Medi Gmbh, Bayreuth, Germany). The Circaid device will be applied with an average pressure of more than 40 mmHg, verified through a BPS (built-in pressure system).
  Interventions: Device: Circaid
- Control arm (No Intervention): No compression

INTERVENTIONS:
Device: Circaid — Circaid is a velcro compression device for the calf (Circaid Juxtalite® Lower Leg; Medi Gmbh, Bayreuth, Germany), thigh and knee (Circaid Juxtafit; Medi Gmbh, Bayreuth, Germany). The Circaid device will be applied with an average pressure of more than 40 mmHg, verified through a BPS (built-in pressure system).
  Arms: Compression arm

SUMMARY:
The objective of the study is to conduct a Bayesian randomized trial comparing non-elastic compression garments applied with high pressure (Circaid group) with no compression (control group) in reducing signs and symptoms in the acute stage of DVT and subsequent postthrombotic syndrome. With a hypothesis that the Circaid group will present a quicker and more marked reduction of pain and leg swelling in the acute stage of DVT, as well as a 20% decrease in the frequency of postthrombotic syndrome within six months from the time of diagnosis of the acute deep vein thrombosis episode.

DETAILED DESCRIPTION:
The pain-relief and edema reduction associated with compressive therapy in patients with acute deep vein thrombosis (DVT) have been poorly documented in randomized controlled trials (RCTs). Compressive therapy is controversial in that it is currently unclear whether or not it might reduce the risk of postthrombotic syndrome (PTS), a chronic disorder identified in 25-50% of patients with a previous diagnosis of deep venous thrombosis. With the recent SOX trial deeming elastic compression stockings to be ineffective in preventing postthrombotic syndrome and with criticisms focused on the difficulty concerning patients' compliance with these devices, alternative methods such as non-elastic compression garments have been considered. Unfortunately, to our knowledge, no trials have investigated these devices applied with a greater pressure than compression stockings in the context of preventing pain and swelling in the acute DVT phase and of late complications (postthrombotic syndrome).

The experimental literature evaluating non-elastic compression garments is primarily focused on venous insufficiency rather than deep vein thrombosis. For example, previous randomized trial patients allocated to non-elastic compression garments presented faster healing rates/week for venous leg ulcers than a group receiving four-layered compression garments. Although this evidence is related to venous insufficiency, there are currently no RCTs exploring the effect of non-elastic compression in preventing postthrombotic syndrome.

Given this gap in the literature, study aimed at conducting a Bayesian randomized trial to assess a non-elastic compression garment (Circaid) versus a control group in patients with acute DVT.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years
* Outpatients with acute deep venous thrombosis of lower extremity
* Symptomatic patients
* Involving femoro-popliteal and / or ilofemoral segment
* Symptoms less than two weeks
* Provoked or unprovoked TVP

Exclusion Criteria:

* History of TVP
* Any allergy to the use of compression material
* Severe arterial occlusive disease
* Patients in whom thrombus removal is planned
* Ankle index <0.5
* Inability to walk
* A life expectancy of less than six months
* Geographic inaccessibility that prevents adequate follow-up with or without assistance
* Thrombolytic therapy outside of this study for the initial treatment of acute DVT.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in pain level using visual analog scale | Baseline visit, after 15 days, one month, six months and 12 months of followup visits.
  Pain level will be registered using a pain visual analog scale (VAS). The pain VAS ranges from 0 (no pain at all) to 10 (very severe pain) and is a self-reported scale where the patient is asked to mark his/her pain level on the line between the two endpoints. A higher score indicates a greater pain intensity.
Change in edema using perimetry (cm) | Baseline visit, after 15 days, one month, six months and 12 months of followup visits.
  The circumference will be measured at two different levels of the foot and at five distinct levels of the leg, using a normal tape measure. No pressure will be applied to these measures to avoid affecting their accuracy. The measurement of the first foot is made five centimeters proximal to the base of the first proximal phalanx of the second toe and the second measurement five centimeters proximal to the first measurement. The measurement of the first leg will be performed five centimeters above the lower edge of the lateral malleolus and then every five centimeters, reaching a total of six to eight measurements, depending on the height of the leg.

SECONDARY OUTCOMES:
Postthrombotic syndrome (PTS) using Ginsberg's criteria | Baseline visit, after 15 days, one month, six months and 12 months of followup visits.
  PTS will be diagnosed following Ginsberg's criteria of ipsilateral pain and swelling of legs at least one month's duration presenting the following characteristics: Worse at the end of the day or with prolonged sitting or standing, and better after a night's rest and with leg elevation.
Postthrombotic syndrome (PTS) using Villalta's scale | Baseline visit, after 15 days, one month, six months and 12 months of followup visits.
  The cumulative incidence and severity of post-thrombotic syndrome (PTS) will be recorded with Villalta's scale. The scale consists of five patient-rated venous symptoms (pain, cramps, heaviness, paresthesia, and pruritis) and six clinician-rated physical signs (pretibial edema, skin induration, hyperpigmentation, pain during calf compression, venous ectasia, and redness) which are each rated on a four-point scale (0=absent, 1=mild, 2=moderate, 3=severe). Points are summed to produce the total score ranging from 0-33. Patients are classified as having PTS if the score is >=5 or if a venous ulcer is present. A score of 5-9 signifies mild disease, 10-14 moderate disease, and ≥15 severe disease.
Quality of life using VEINES-QOL/Sym questionnaire | Baseline visit and at one, six and 12 months of followup visits.
  VEnous INsufficiency Epidemiological and Economic Study- Quality of Life/ Symptoms (VEINES-QOL/Sym) is a 26-item patient-reported questionnaire measuring the impact of deep venous thrombosis on symptoms and quality of life. Out of two summary scores, the VEINES-QOL summary score (25 items) provides an estimate of the overall impact of deep venous thrombosis on the patient's quality of life and the VEINES-Sym summary score (10 items) measures symptom severity. This includes nine venous symptoms (heavy legs, aching legs, swelling, night cramps, heat or burning sensation, restless legs, throbbing, itching, tingling sensation), rated on a five-point Likert scale of frequency (every day, several times a week, about once a week, less than once a week, never), and leg pain rated on a six-point scale of intensity (very severe, severe, moderate, mild, very mild, none). For both scales, high scores indicate better outcomes.
Quality of life using PROMIS Global-10 | Baseline visit and at one, six and 12 months of followup visits.
  PROMIS-10 assesses general domains of health and functioning including overall physical health, mental health, social health, pain, fatigue, and overall perceived quality of life.
Physical activity using Global Physical Activity Questionnaire | Baseline visit and at one, six and 12 months of followup visits.
  Global Physical Activity Questionnaire (GPAQ) developed by WHO collects information on physical activity participation in three settings (or domains) as well as sedentary behavior, comprising 16 questions (P1-P16). The domains are: Activity at work; Travel to and from places; Recreational activities. Metabolic Equivalents (MET) are commonly used to express the intensity of physical activities, and are also used for the analysis of GPAQ data. MET is the ratio of a person's working metabolic rate relative to the resting metabolic rate. One MET is defined as the energy cost of sitting quietly, and is equivalent to a caloric consumption of 1 kcal/kg/hour. When calculating a person's overall energy expenditure using GPAQ data, 4 METs get assigned to the time spent in moderate activities, and 8 METs to the time spent in vigorous activities.

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Matta, MD, Principal Investigator — Pró Circulação®
Locations (18):
- Brazil (18):
  - Instituto de Ensino e Treinamento em Saúde Vascular da Bahia, Salvador, Estado de Bahia
  - Angiodiagnóstico - Instituto de Doenças Venosas e Linfáticas de Goiânia/Go, Goiânia, Goiás
  - Clínica Médica Longevittá, Cuiabá, Mount
  - Instituto de Cirurgia Vascular e Angiologia de Cascavel/PR, Cascavel, Paraná
  - Hospital Erasto Gaertner, Curitiba, Paraná
  - Hospital Santa Casa de Curitiba, Curitiba, Paraná
  - NICEP - Núcleo Integrado de Cirurgia Vascular e Pesquisa, Curitiba, Paraná
  - Sociedade Evangélica Beneficente de Curitiba, Curitiba, Paraná
  - Flebocurso, Londrina, Paraná
  - Hospital dos Servidores do Estado do Pernambuco, Recife, Pernambuco
  - Angio Vascular Hospital LTDA, Natal, Rio Grande do Norte
  - Centro: Serviço de Cirurgia Vascular HSLPUCRS, Porto Alegre, Rio Grande do Sul
  - Clínica vascular MDC Sociedade Simples ME, Porto Alegre, Rio Grande do Sul
  - Pró Saúde Clínica Médica, Tubarão, Santa Catarina
  - Pró Circulação® - Clinic of Angiology and Vascular Surgery, Xanxerê, Santa Catarina
  - Clínica Dr. Alexandre Reis EIRELI, Santos, São Paulo
  - CIP - Fundação Faculdade de Medicina de São José do Rio Preto, São José do Rio Preto, São Paulo
  - SAMAR Serviços Médicos, São Paulo, São Paulo

REFERENCES:
- See also: Circaid, a non-elastic compression garment — https://www.medi.de/en/products/highlights/circaid/